CLINICAL TRIAL: NCT02410083
Title: Multicenter, Randomized, Open Study, Investigator-initiated Trial for Comparison of Eight Weeks Efficacy and Tolerability of Clopirin and Clopidogrel With Aspirin in Korean Patients With Post-Percutaneous Coronary Artery Intervention
Brief Title: Trial to Assess the Efficacy of Combination Formula of Aspirin Plus Clopidogrel in Patients With Coronary Stent
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JP_CLN_01
Record Dates: First submitted 2015-03-19; First posted 2015-04-07 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2015-03

CONDITIONS: ANEURYSM CORONARY ARTERY
MeSH Terms: conditions — Coronary Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Clopirin 1 (Experimental): Clopirin single-administration. Before this clinical trial Clopidogrel/Aspirin co-administration.
  Interventions: Drug: Clopirin 1
- Clopidogrel/Aspirin co-administration 1 (Active Comparator): Clopidogrel-aspirin co-administration. Before this clinical trialClopidogrel/Aspirin co-administration.
  Interventions: Drug: Clopidogrel-Aspirin(co-administration) 1
- Clopirin 2 (Experimental): Clopirin single-administration. Before this clinical trial Aspirin single-administration.
  Interventions: Drug: Clopirin 2
- Clopidogrel/Aspirin co-administration 2 (Active Comparator): Clopidogrel-aspirin-co-administration. Before this clinical trial Aspirin single-administration.
  Interventions: Drug: Clopidogrel-Aspirin(co-administration) 2

INTERVENTIONS:
Drug: Clopirin 1
  Arms: Clopirin 1
Drug: Clopidogrel-Aspirin(co-administration) 1
  Arms: Clopidogrel/Aspirin co-administration 1
Drug: Clopirin 2
  Arms: Clopirin 2
Drug: Clopidogrel-Aspirin(co-administration) 2
  Arms: Clopidogrel/Aspirin co-administration 2

SUMMARY:
The purpose of this study in to evaluate efficacy and tolerability of Clopirin and clopidogrel with aspirin in Korean Patients with post-percutaneous coronary artery intervention.

ELIGIBILITY:
Inclusion Criteria:

* Over 3 months, the patient who were the administration of aspirin or the co-administration of clopidogrel-aspirin coronary artery patients after treated with Percutaneous Coronary Intervention(PCI) that have safety progress.
* Korean men and women between the age of 20 and 85
* Patients who understand the study requirements, are willing to comply with all study procedures and have provided written informed consent.

Exclusion Criteria:

* Patients who were not treated with PCI or intended to treat with PCI but failed.
* Patients who were taking or had taken other antiplatelet or anticoagulant for more than 2 weeks within the prior 30 days.
* Patients who had a history of alcohol abuse or intoxication.
* Patients who had hypersensitivity to clopidogrel or aspirin.
* Patients who had severe hepatic dysfunction aspartate aminotransferase(AST) or alanine aminotransferase(ALT) > 3 times upper normal reference values.
* Patients who had blood coagulation disorders, uncontrolled severe hypertension, active bleeding, or history of severe bleeding, such as intracranial hemorrhage or ulcer bleeding - surgery within 48hr, platelet counts below 50,000/mm3 in laboratory tests.
* Patients who were pregnant, breastfeeding.
* Patients who were not using effective methods of contraception. (proper contraception : hormonal contraception, condom, intrauterine device, spermicide)
* Patients who medically, psychologically had investigational product administration's prohibition.
* Patients who were not participated in this clinical trial decided by other investigators.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
% inhibition =△Purinergic receptor, G-protein coupled, 12 Reaction Units(PRU)/ Pretreatment PRU | 8 weeks

SECONDARY OUTCOMES:
△ PRU = Post treatment PRU - Pre treatment PRU | 8 weeks
△ ARU = Post treatment Aspirin resistance unit(ARU) - Pre treatment ARU | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-soo Kim, Professor, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No